CLINICAL TRIAL: NCT03040791
Title: Nivolumab in Prostate Cancer With DNA Repair Defects (ImmunoProst Trial)
Acronym: ImmunoProst
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64121317.4.1001.5330
Record Dates: First submitted 2017-01-27; First posted 2017-02-02 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a Phase II, two-stage, multi-center, single-arm, and open-label trial of Nivolumab (BMS-936558) in patients with mCRPC who have progressed to a taxane-based chemotherapy regimen previously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab (Experimental): All patients will receive Nivolumab 240 mg every 14 days until progression or unacceptable toxicity
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab
  Other Names: BMS-936558

SUMMARY:
Prostate Cancer (PC) is the most frequent cancer in men, accounting for 21% of new cases of cancer in men in the United States. Among the four most incident tumors (breast, lung and colorectal cancer); prostate cancer is the only that does not have any predictive biomarker to guide the treatment. Even though the molecular heterogeneity of PC is well-documented, treatment has not been molecularly stratified and the need for genetic prognostic and predictive markers is critical.

DNA repair defects (DRD), mainly in the Homologous Recombination (HR) pathway (such as BRCA1, BRCA2, ATM and CHEK2) are emerging as potential biomarkers in prostate cancer. It is well known BRCA1 and BRCA2 carriers have better Progression-Free Survival (PFS) and Overall Survival (OS) than non-carriers in ovarian cancer. Differently than ovarian tumors that BRCA mutations provides a good prognosis, PC patients who harbor HR defects have a higher Gleason score 6, an increased risk of recurrence and poor prognosis. The predictive role of DRD in PC was demonstrated in a recent trial using Olaparib, a PARP inhibitor, in DRD carriers. This trial showed 88% of response rate with Olaparib, a PARP inhibitor that acts in HR pathway by synthetic lethality.

Recent data demonstrated important association between HR deficient high-grade serous ovarian cancer (HGSOC), high neoantigen load and high expression of PD-1/PD-L1 compared with HR proficient HGSOCs 10. This study showed that BRCA1 and BRCA2 mutations increase the number of tumor-infiltrating lymphocytes (TILs) and confer a better prognosis. The unprecedented success of immunotherapy in malignant disorders has provided evidence that the patient's immune system can be improved to attack established tumors, mainly melanoma, non-small cell lung cancer and kidney cancer. A high mutational burden increases the likelihood of the development of specific neoepitopes that would confer clinical benefit from CTLA-4 and PD-1 blockade.

These data showed that specific DNA repair defects increase the mutational burden, the expression of PD-1/PD-L1 and TILs; and could improve the response to immunotherapy in cancer. This rationale was already tested in a trial that evaluated the PD-1 checkpoint inhibitor Pembrolizumab in mismatch-repair deficient patients, a kind of DNA repair defect by definition. This important trial showed that this DRD predicted clinical benefit of immune checkpoint blockade in many types of cancer, especially colorectal cancer.

DETAILED DESCRIPTION:
This is a Phase II, two-stage, multi-center, single-arm, and open-label trial of Nivolumab (BMS-936558) in patients with metastatic castration-resistant prostate cancer (mCRPC) who have progressed to a taxane-based chemotherapy regimen previously. Eligible patients must have ECOG 0-2 and material for biomarker analysis. Prior enzalutamide, abiraterone and cabazitaxel are permitted but not necessary to enrollment. The germline and somatic DRD (BRCA1, BRCA2, ATM, PTEN, CHEK2, RAD51C, RAD51D, PALB2, MLH1, MSH2, MSH6, PMS2.) will be assessed by T-NGS of metastatic sites or by liquid biopsy. The primary endpoint is PSA 50 response rate (PSA50, following the Prostate Cancer Working Group 3 criteria). The trial will meet its endpoint if ≥ 3/29 men achieve a PSA50 response. The secondary endpoints will include progression-free survival (PFS), overall survival, radiologic PFS, PSA response rate at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate with tumor tissue available for molecular analyses. If archival tissue for biomarker analysis is not available then the patient must be willing to have a further biopsy to obtain tumor tissue for histological diagnosis.
2. Metastatic Castrate-resistant prostate cancer (mCRPC), defined by:

   * Disease progression despite androgen deprivation therapy (ADT) and may present as either a continuous rise in serum prostate-specific antigen (PSA) levels, the progression of pre-existing disease, and/or the appearance of new metastases.
   * Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If the patient is being treated with GnRH or LHRH agonists or antagonists (patient who have not undergone orchiectomy), this therapy should be maintained.
3. Documented prostate cancer progression, during treatment with Docetaxel, as assessed by the investigator with one of the following:

   * PSA progression is defined according the PCWG3 criteria: PSA increase, that is ≥ 50% and ≥ 2 ng/mL above the nadir, and which is confirmed by a second value ≥ 3 weeks later (confirmed the rising trend).
   * Radiographic progression of visceral lesions or soft tissue disease by modified RECIST 1.1 criteria.
   * Progression of bone metastasis is defined according the Appendix B: Prostate Cancer Clinical Trials Working Group 3 (Adapted) two or more documented new bone lesions on a bone scan with or without PSA progression. Confirmation of ambiguous results by other imaging modalities (eg, CT or MRI) is obligatory. If Docetaxel chemotherapy is used more than once, this will be considered as one regimen.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 Appendix A: Performance Status Criteria
5. Life expectancy > 24 weeks.
6. Age ≥ 18 years
7. At least 28 days since the completion of any prior anti-cancer therapy (except for LHRH agonists or antagonists), including chemotherapy (taxane-based). Additionally, clinically relevant treatment toxicities should have resolved to grade 1 or less prior to start study treatment.
8. For hormonal treatment must be followed the guideline below:

   * No antiandrogens are allowed during the study period. The use of antiandrogens before study entry is permitted, but at least 28 days since the completion of prior antiandrogen are required (washout period).
   * Corticosteroids dose > Prednisolone 10 mg/day (or equivalent) are allowed only if clinically indicated for medical conditions. At least 28 days since the completion of prior corticotherapy are required (washout period).
9. Agreeable to have all the biomarker studies including the fresh tumor biopsies if needed.
10. Patients must have adequate organ function within 1 weeks prior enrollment to and evidenced by:

    * Hemoglobin ≥ 9.0 g/dL
    * WBC > 2.000/mm3
    * Absolute neutrophil count ≥ 1.500/mm3
    * Platelet count ≥ 100.000/mm3
    * Creatinine Clearance ≥ 30 mL/min. Creatinine Clearance (CrCl) must be calculated at screening using the Cockcroft-Gault formula:
    * Bilirubin < 3 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome.
    * Aspartate transaminase (AST) (SGOT) < 3.0 x ULN.
    * Alanine transaminase (ALT) (SGPT) < 3.0 x ULN.
    * No cardiac disease defined by as active angina, symptomatic congestive heart failure, or myocardial infarction within previous six months.

Exclusion Criteria:

* Patients with any active known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, controlled autoimmune hypothyroidism, psoriasis not requiring systemic treatment, or other conditions under control are permitted to enroll.
* Patients with conditions that needs systemic corticosteroids dose > Prednisolone 10 mg/day (or equivalent) or other immunosuppressive medications within 28 days prior to the first dose of study drug. Inhaled steroids are permitted if necessary.
* Patients with any known active chronic liver disease.
* Patients who have prior history of malignancy treated with curative intention in the past 2 years with the exception of basal cell carcinoma and squamous cell carcinoma of the skin, which were allowed in any case. Patients with other malignancies that do not fulfill the prior criteria could be considered for recruitment if they do not represent a competitive cause of death and have a low potential to progress to metastatic progression. Patients in this condition may be enrolled in the trial if approved after review by principal investigator.
* Known history of testing positive for human immunodeficiency virus (HIV), known acquired immunodeficiency syndrome (AIDS), or any positive test for hepatitis B or hepatitis C virus representing acute or chronic disease.
* Preceding treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Major surgery less than 28 days prior to the first dose of study drug.
* Radiation therapy less than 14 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
PSA response rate | through study completion, an average of 1 year
  PSA partial response is defined as a ≥ 50% decline in PSA from cycle 1 day 1 (baseline) PSA value. This PSA decline must be confirmed as sustained by a second PSA value obtained ≥ 3 weeks later.

SECONDARY OUTCOMES:
Time to PSA progression | through study completion, an average of 1 year
PSA Response Rate at 6 and 12 months | through study completion, an average of 1 year
Radiological progression-free survival (rPFS) | through study completion, an average of 1 year
Time to Radiographic Progression | through study completion, an average of 1 year
Progression free survival (PFS) | through study completion, an average of 1 year
Overall survival | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Isaacsson, MD, Principal Investigator — Hospital Moinhos de Vento
Locations (2):
- Brazil (2):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of study For 1 year
Access Criteria: RedCap / Excel